CLINICAL TRIAL: NCT07150858
Title: Comparison Between Erythropoietin-enhanced Albumin Platelet-rich Fibrin and Albumin Platelet-rich Fibrin in Transcrestal Sinus Lifting With Simultaneous Implant Placement
Brief Title: Erythropoietin - Albumin Platelet-rich Fibrin in Transcrestal Sinus Lifting With Simultaneous Implant Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1073-5/2025
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Sinus Lifting
Keywords: Transcrestal sinus lifting, erythropoitein, albumin PRF, Peizo electric device, Dental implants, CBCT.
MeSH Terms: interventions — Erythropoietin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erythropoietin and albumin PRF gel (Experimental)
  Interventions: Other: Erythropoietin and albumin PRF gel + implant placement
- albumin PRF gel (Active Comparator)
  Interventions: Other: Albumin PRF gel +implant placement

INTERVENTIONS:
Other: Erythropoietin and albumin PRF gel + implant placement — This group will be treated by transcrestal sinus lifting with erythropoietin and albumin PRF gel with simultaneous implant placement.
  Arms: Erythropoietin and albumin PRF gel
Other: Albumin PRF gel +implant placement — This group (the Control group) will be treated with transcrestal sinus lifting using albumin PRF gel, with simultaneous implant placement.
  Arms: albumin PRF gel

SUMMARY:
Background: Dental implant therapy in the posterior maxilla may be difficult owing to limited bone height after dental extraction with sinus pneumatization. Several approaches for sinus floor elevation have been documented, and hence trans crestal sinus lifting with albumin platelet rich plasma.

Aim of the study: To compare between erythropoietin and albumin platelet rich fibrin transcrestal sinus lifting versus albumin platelet rich fibrin transcrestal sinus lifting using piezoelectric device in patients with atrophic maxilla.

Methods: This study will be carried out as a randomized

ELIGIBILITY:
Inclusion Criteria:

* Residual bone height not less than 5 mm measured from crestal bone to sinus floor.
* Both genders.
* Good oral hygiene
* No previous surgery or radiation treatment on the maxillary sinus

Exclusion Criteria:

* Recent radiation therapy in maxilla.
* Uncontrolled systemic diseases such as diabetes mellitus.
* Heavy smoker (those who smoke ≥ 25 cigarettes a day).
* Alcohol abuse.
* Patient on anticoagulant drug
* Severe allergic rhinitis.
* Tumor or large cyst in the maxillary sinus.
* Oroantral fistula.
* Presence of acute or chronic sinus pathoses or sinus membrane perforation.(

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2026-07-25 (Estimated); Study Completion 2026-07-25 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores | up to 14 days
  pain will be assessed through a 10 point visual analogue scale (VAS). (0-1=none, 2-4=mild, 5-7=moderate, 8-10=severe).
Change in edema | up to 14 days
  Edema will be assessed as follows:
  1. None (no swelling)
  2. Mild (intraoral swelling confined to the surgical field)
  3. Moderate (extra oral swelling in the surgical zone)
  4. Severe (extraoral swelling spreading beyond the surgical zone)
Change in implant stability | immediate and 4 months
  implant stability will be assessed using ostell device

SECONDARY OUTCOMES:
Change in bone gain | baseline and 4 months
  amount of sinus bone gain (SBG) which equals implant protrusion length (IPL) added to Peri-implant sinus bone level (PSBL) which is the distance between the apex of the implant and sinus bone level
Change in bone density | baseline and 4 months
  it will be assessed using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt